CLINICAL TRIAL: NCT01247155
Title: First Postoperative Day Review After Uneventful Phacoemulsification
Status: Completed | Type: Observational
Sponsor: Veroia General Hospital (Other)
Other Study IDs: 9151
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2009-04

CONDITIONS: Phacoemulsification; Complications; BCVA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- first day review
- non-first day review

SUMMARY:
The purpose of this randomized trial was to examine the value of the review on the first postoperative day after uneventful phacoemulsification cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

Exclusion criteria were the following:

i) intra-operative complications, such as posterior capsule rupture, vitreous loss, lost nucleus, zonule dehiscence and wound leak,

ii) inadequate social support for overnight care at home,

iii) severely limited visual potential in the fellow eye,

iv) uveitis or ocular trauma,

v) severe systemic diseases limiting activity,

vi) patients with learning disability or dementia.

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: 291 consecutive patients who underwent uneventful phacoemulsification cataract surgery were randomized into two groups: i) Next day review (NDR group, n=146) and ii) No next day review (NNDR group, n=145).
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Veroia, Véroia, Imathia, Greece

REFERENCES:
- [Derived] Chatziralli IP, Sergentanis TN, Kanonidou E, Papazisis L. First postoperative day review after uneventful phacoemulsification cataract surgery: is it necessary? BMC Res Notes. 2012 Jun 27;5:333. doi: 10.1186/1756-0500-5-333. PMID 22738668